CLINICAL TRIAL: NCT03658746
Title: Efficacies of Antimicrobial Susceptibility-Guided Versus Empirical Therapy for Rescue Treatment of Helicobacter Pylori Infection-A Randomized Clinical Trial
Brief Title: Efficacies of Antimicrobial Susceptibility-Guided Versus Empirical Therapy for Rescue Treatment of Helicobacter Pylori Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Xiuli Zuo, director of Qilu Hospital gastroenterology department, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018SDU-QILU-G003
Record Dates: First submitted 2018-09-02; First posted 2018-09-05 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Helicobacter Pylori Infection
Keywords: Antimicrobial Susceptibility Testing; Rescue Therapy
MeSH Terms: interventions — Clarithromycin; Metronidazole; Tinidazole; Levofloxacin; Furazolidone; Tetracycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antimicrobial susceptibility guided therapy (Experimental): Patients in this group will receive a 14-day quadruple therapy for helicobacter pylori eradication. The regimen contains one proton pump inhibitor, colloidal bismuth pectin, and two sensitive antibiotics determined by antimicrobial susceptibility test. The susceptibility of amoxicillin, clarithromycin, metronidazole, tinidazole, levofloxacin, furazolidone and tetracycline will be evaluated.
  Drugs: 1.one proton pump inhibitor: rabeprazole 10mg bid for 14d, 2.Colloidal Bismuth Pectin 200mg bid for 14d, 3.two sensitive antibiotics: amoxicillin 1000mg bid for 14d, clarithromycin 500mg bid for 14d, metronidazole 500mg tid for 14d, tinidazole 500mg tid for 14d, levofloxacin 500mg qd for 14d, furazolidone 100mg bid for 14d, tetracycline 500mg qid for 14d.
  Interventions: Drug: two sensitive antibiotics(amoxicillin, clarithromycin, metronidazole, tinidazole, levofloxacin, furazolidone and tetracycline); Drug: one proton pump inhibitor, colloidal bismuth pectin
- Empirical therapy according to medication history (Active Comparator): Patients in this group will receive a 14-day quadruple therapy based on personal medication history for helicobacter pylori eradication. The regimen contains one proton pump inhibitor, Colloidal Bismuth Pectin and two antibiotics chosen according to medication history. If the patient hasn't been treated with levofloxacin in the previous eradication regimen, he will be treated with amoxicillin and levofloxacin. Otherwise, he will be treated with amoxicillin and furazolidone.
  Drugs: 1.one proton pump inhibitor: rabeprazole 10mg bid for 14d 2.Colloidal Bismuth Pectin 200mg bid for 14d 3.two antibiotics based on personal medication history: amoxicillin 1000mg bid and levofloxacin 500mg qd for 14d, amoxicillin 1000mg bid and furazolidone 100mg bid for 14d.
  Interventions: Drug: one proton pump inhibitor, colloidal bismuth pectin; Drug: two antibiotics based on personal medication history(amoxicillin,levofloxacin, furazolidone)

INTERVENTIONS:
Drug: two sensitive antibiotics(amoxicillin, clarithromycin, metronidazole, tinidazole, levofloxacin, furazolidone and tetracycline) — Patients will receive a 14-day quadruple therapy for the H.pylori eradication. The regimen contains one proton pump inhibitor, colloidal bismuth pectin and two sensitive antibiotics determined by antimicrobial susceptibility test. The susceptibility of amoxicillin, clarithromycin, metronidazole, tinidazole, levofloxacin, furazolidone and tetracycline will be evaluated.
  Arms: Antimicrobial susceptibility guided therapy
Drug: one proton pump inhibitor, colloidal bismuth pectin — All patients need these two drugs.
Drug: two antibiotics based on personal medication history(amoxicillin,levofloxacin, furazolidone) — Patients will receive a 14-day quadruple therapy according to personal medication history for helicobacter pylori eradication. The regimen contains one proton pump inhibitor, Colloidal Bismuth Pectin and two antibiotics based on personal medication history. If the patient hasn't been treated with levofloxacin previously, he will be treated with amoxicillin and levofloxacin. Otherwise, he will be treated with amoxicillin and furazolidone.
  Arms: Empirical therapy according to medication history

SUMMARY:
The purpose of this study is to assess efficacy of 14-day antimicrobial susceptibility test guided quadruple therapy for the rescue treatment of Helicobacter pylori infection, then comparing it with 14-day empirical therapy according to personal medication history.

DETAILED DESCRIPTION:
Helicobacter pylori(H.pylori), which infects about 50% of the global population, has been classified as the first risk factor of gastric cancer. Strong evidence supports that H.pylori eradication is an effective approach to reduce the incidence of those pathological processes. Antimicrobial susceptibility test can pick out sensitive drugs to kill H.pylori, and reduce secondary drug resistance. However, there is a lack of high quality RCT to evaluate its efficacy in the rescue treatment of Helicobacter infection.

The investigator's study aims to assess the efficacy of 14-day antimicrobial susceptibility test guided quadruple therapy for the rescue treatment of Helicobacter pylori infection. Then, comparing this regimen with 14-day empirical therapy according to personal medication history to tell which one is better in clinic practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-70 with persistent Helicobacter pylori infection.
* Patients with previous Helicobacter pylori eradication therapy for one or two times.

Exclusion Criteria:

* Patients unable or unwilling to receive gastroscopy.
* Patients treated with Histamine-receptor antagonist, proton pump inhibitor, bismuth and antibiotics in the previous 4 weeks.
* Patients with gastrectomy, acute gastrointestinal bleeding and advanced gastric cancer.
* Patients with known or suspected allergy to study medications.
* Currently pregnant or lactating.
* Inability to provide informed consent and other situations that could interfere with the examination or therapeutic protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 420 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Eradication rates | 6 months
  Both intention to treat(ITT) and per-protocol(PP) analyses will be used for the assessment of the eradication rates of Helicobacter pylori infection. The ITT analysis includes all randomly assigned patients who take at least one dose of the study medications. The PP analysis is limited to patients who take over 90% of the study medications and complete follow-up.

SECONDARY OUTCOMES:
The rates of adverse events happening | 6 months
  Common adverse events will be measured using a 8-point Likert scale, and patients rate their symptoms from 0 (none) to 8 (severe) during the treatment process.
The rates of improving dyspepsia symptoms after helicobacter pylori eradication. | 6 months
  Dyspepsia symptoms will also be measured using a 8-point Likert scale.be compared. Common adverse events will be measured using a 8-point Likert scale. Patients rate their symptoms from 0 (none) to 8 (severe) before and after the treatment process.
The rates of good compliance. | 6 months
  Patients taken over 90% of drugs are considered to have a good compliance.

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Zuo, MD,PhD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu hosipital, Jinan, Shandong, China